CLINICAL TRIAL: NCT06629324
Title: Evaluation of the Efficacy of Autologous Bone Marrow-Derived Mononuclear Cell Transplantation in the Treatment of Cerebral Palsy Due to Brain Hypoxia: A Phase II Randomized Clinical Trial
Brief Title: Evaluating Bone Marrow Cell Transplant for Treating Cerebral Palsy From Brain Hypoxia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISC-22.72
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BM MNC transplantation and Rehabilitation (Active Comparator): Patients in group A will receive two autologous BM MNC administrations at baseline and 6 months ± 21 days (T6)
  Interventions: Biological: Autologous Bone Marrow Mononuclear Cell Transfusion; Other: Rehabilitation
- Placebo with Rehabilitation, then BM MNC transplantation (Placebo Comparator): Group B will receive BM MNCs at 9 months ± 21 days (T9) and 15 months ± 21 days (T15), with outcomes evaluated at 18 months ± 21 days (T18) compared to baseline.
  Interventions: Biological: Autologous Bone Marrow Mononuclear Cell Transfusion; Other: Rehabilitation

INTERVENTIONS:
Biological: Autologous Bone Marrow Mononuclear Cell Transfusion — Bone marrow was collected under general anesthesia from both anterior superior iliac crests, taking 15-20 minutes, with a maximum volume of 350 mL for older children. Mononuclear cells were isolated using Ficoll density gradient centrifugation and prepared for infusion. The infusion, performed in the L4-L5 spinal space, lasted about 30 minutes at a rate of 20 mL per hour. Cerebrospinal fluid (CSF) was withdrawn before infusion, with the amount based on the child's weight. Patients received Rocephin for infection prevention and pain relief with alternating doses of Ibuprofen and Efferalgan for 2 days post-procedure. Seduxen was given once on the first night after bone marrow collection.
Other: Rehabilitation — Rehabilitation methods involve various therapies tailored to the patient's mobility level. (1) Physical therapy focuses on exercises to control the head, neck, and trunk, manage muscle tone, and reduce spasticity. Patients gradually practice essential movements like rolling, sitting, crawling, standing, and walking, aligned with developmental milestones. (2) Occupational therapy aims to enhance fine motor skills and daily activities. Through hand function exercises, patients improve upper limb functionality, strengthen their ability to grasp and hold objects and refine coordination between both hands and hand-eye coordination. (3) Speech therapy improves communication, cognitive abilities, and chewing and swallowing functions. Specific exercises target lip and mouth movements, helping patients express and understand language better. Additionally, there are activities to strengthen jaw and facial muscles, which are essential for improving chewing and swallowing abilities.

SUMMARY:
This clinical trial aims to evaluate the effectiveness of autologous bone marrow mononuclear cell transfusion in treating cerebral palsy caused by cerebral hypoxia.

The key questions the study seeks to answer are:

* What is the safety profile in terms of adverse events (AE) and serious adverse events (SAE) observed over the 9 months following the first transplantation?
* How does autologous bone marrow mononuclear cell (BM MNC) transplantation impact the gross motor function (GMFM-88) scores and Gross Motor Function Classification System (GMFCS) scores in children with cerebral palsy?
* How does autologous BM MNC transplantation influence muscle tone (Modified Ashworth Scale score) and hand motor function (MACS/Mini-MACS scale) in children with cerebral palsy, 9 months post the initial transplantation?

Fifty-eight selected patients, aged 1 to 10 years and diagnosed with spastic cerebral palsy due to brain hypoxia, will be randomly divided into two groups:

* Group A: will receive two BM MNC infusions with the first at baseline and the second at 6 months ± 21 days (T6) via the spinal route.
* Group B: will serve as the control group for the first 9 months. During this period, patients will not receive cell transplantation but will undergo a similar rehabilitation and medication regimen as Group A. After 9 months, Group B will receive two BM MNC infusions: the first at 9 months ± 21 days (T9) and the second at 15 months ± 21 days (T15) via the spinal route, with a follow-up at 18 months ± 21 days (T18) compared to baseline.
* Both groups: will undergo rehabilitation for 10 days per month, three times, either at rehabilitation centers or performed by a rehabilitation technician at home. After this period, continued training will be conducted by family members. The combined medication regimen will include muscle relaxants (if muscle spasticity is present), vitamins, and neuroprotective drugs (Piracetam).

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is one of the most common causes of motor disability in children, significantly affecting their quality of life (QOL). Children with CP often face various challenges, including motor, sensory, and communication difficulties [1]. Recent studies suggest that autologous bone marrow-derived mononuclear cells (BM MNCs) show promise in improving motor function and reducing muscle spasticity in CP children [2, 3, 4]. The effects of BM MNC transplantation on the quality of life in CP children and their families remain understudied, despite improvements in motor function being reported.

Our Phase I study evaluated the safety and effects of autologous BM MNCs on the improvement of gross motor function and muscle tone in children with CP. This Phase II randomized clinical trial aims to evaluate the efficacy of autologous BM MNCs in children with CP at Vinmec International Hospital, Hanoi, Vietnam, from October 2024 to January 2027 [5]. The inclusion criteria are: (1) aged 1 to 10 years and of either sex; (2) having a Gross Motor Function Classification System (GMFCS) score ranging from level II to level V; and (3) spastic cerebral palsy due to cerebral hypoxia. Patients will be excluded if they have coagulation disorders; suffer from severe health conditions such as exhaustion, heart, lung, liver, or kidney failure, or active infections; have spinal injuries that prevent the administration of intrathecal injections; are diagnosed with cancer; test positive for HIV or have active viral hepatitis; or have hemoglobin levels below 110 g/L.

In total, 58 patients were randomly assigned to two groups. Randomization allocation was conducted using a random number table, and the ratio of participants in each group was 1:1. Group A will receive two BM MNC administrations: the first at baseline and the second at 6 months ± 21 days (T6) via intrathecal injection. Concomitantly, the CT group will undergo a 10-day-per-month rehabilitation program for 3 months, either at rehabilitation centers or with at-home therapy, followed by exercises managed by family members. Group B will serve as the control group for the first 9 months, receiving rehabilitation and medications similar to Group A but without BM MNC therapy. After 9 months, Group B will receive BM MNCs at 9 months ± 21 days (T9) and 15 months ± 21 days (T15), with outcomes evaluated at 18 months ± 21 days (T18) compared to baseline.

Bone marrow was collected under general anesthesia from both anterior superior iliac crests, taking 15-20 minutes, with a maximum volume of 350 mL for older children. Mononuclear cells were isolated using Ficoll density gradient centrifugation and prepared for infusion. The infusion, performed in the L4-L5 spinal space, lasted about 30 minutes at a rate of 20 mL per hour. Cerebrospinal fluid (CSF) was withdrawn before infusion, with the amount based on the child's weight. Patients received Rocephin for infection prevention and pain relief with alternating doses of Ibuprofen and Efferalgan for 2 days post-procedure. Seduxen was given once on the first night after bone marrow collection. The rehabilitation program included exercises for head and body control, muscle tone management, and facilitated movements based on developmental milestones. Occupational therapy focused on improving hand function and daily activities, while speech therapy addressed communication, comprehension, and chewing/swallowing abilities.

The safety of the therapy will be assessed by monitoring the frequency and severity of adverse events (AEs) and serious adverse events (SAEs). SAEs include events leading to death, life-threatening conditions, hospitalizations or prolonged hospital stays, significant or permanent disabilities, and congenital abnormalities or birth defects. Efficacy will be evaluated based on changes in gross motor function 9 months after the first BM MNC transplant. This will involve the GMFM-88 scale to assess gross motor function, the GMFCS scale to classify motor function severity, and the Mini-MACs (for children aged 1-4) and MACs (for children aged 4-18) scales to measure hand function. Additionally, muscle tone changes will be measured using the Modified Ashworth Scale 9 months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age from 1 to 10 years, both genders;
* Gross Motor Function Classification System (GMFCS): levels II to V;
* Spastic cerebral palsy due to brain hypoxia.

Exclusion Criteria:

* Coagulation disorders;
* Severe health conditions such as cachexia, heart failure, lung, liver, or kidney failure; or active infections;
* Spinal injuries prevent the placement of a catheter through the spinal cavity;
* Cancer;
* HIV positive, active viral hepatitis;
* Hemoglobin below 110 g/L.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events and Serious adverse events | Up to 9 months for Group A and 18 months for Group B during the study.
  The incidence of adverse events or serious adverse events following transplantation includes events leading to death, life-threatening events, events requiring hospitalization or prolonging hospital stay, events resulting in significant or permanent disability, and events causing birth defects in newborns.
Gross Motor Function Measure-88 (GMFM-88) | Group A: Baseline; 3 months (T3±21 days); 6 months (T6±21 days); 9 months (T9±21 days)/ Group B: Baseline; 3 months (T3±21 days); 6 months (T6±21 days); 9 months (T9±21 days); 12 months (T12±21 days); 15 months (T15±21 days); 18 months (T18±21 days).
  Evaluate the effectiveness of umbilical cord blood stem cell transplantation in children with cerebral palsy based on changes in gross motor function score after the first cell transplantation.
Gross Motor Function Classification System (GMFCS) | Group A: Baseline; 3 months (T3±21 days); 6 months (T6±21 days); 9 months (T9±21 days). Group B: Baseline; 3 months (T3±21 days); 6 months (T6±21 days); 9 months (T9±21 days); 12 months (T12±21 days); 15 months (T15±21 days); 18 months (T18±21 days).
  This tool will be used to classify the severity of motor function impairment in children with cerebral palsy.
The Mini-Manual Ability Classification System (Mini-MACS) and Manual Ability Classification System (MACS) | Group A: Baseline; 3 months (T3±21 days); 6 months (T6±21 days); 9 months (T9±21 days). Group B: Baseline; 3 months (T3±21 days); 6 months (T6±21 days); 9 months (T9±21 days); 12 months (T12±21 days); 15 months (T15±21 days); 18 months (T18±21 days).
  Hand function after the first cell transplantation: Mini-MACS (Manual Ability Classification System) for children aged 1 to 4 years, and MACS for children aged over 4 to 18 years.
Modified Ashworth Scale | Group A: Baseline; 3 months (T3±21 days); 6 months (T6±21 days); 9 months (T9±21 days). Group B: Baseline; 3 months (T3±21 days); 6 months (T6±21 days); 9 months (T9±21 days); 12 months (T12±21 days); 15 months (T15±21 days); 18 months (T18±21 days).
  Change in muscle tone after the first cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Liem T Nguyen, MD., PhD, Principal Investigator — Vinmec Research Insitute of Stem Cell and Gene Technology
Locations (2):
- Vietnam (2):
  - Vinmec research Institute and Gene Technology, Hanoi
  - Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi

IPD SHARING:
Plan to Share IPD: No